CLINICAL TRIAL: NCT00155285
Title: Integrated Evaluating the Infant Complex Congenital Heart Disease by Multidetector(16)Spiral Computed Tomography
Brief Title: Evaluating the Infant Complex Congenital Heart Disease by Multidetector Computed Tomography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 9361700485
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-10-20 (Estimated); Status verified 2003-04

CONDITIONS: Heart Diseases
Keywords: heart diseases; congenital
MeSH Terms: conditions — Heart Diseases

INTERVENTIONS:
Procedure: computed tomography

SUMMARY:
To test the ability of multi-detector spiral CT in evalting the infant complex congenital heart disease.

DETAILED DESCRIPTION:
To test the ability of multi-detector spiral CT in evalting the infant complex congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

complex congenital heart disease

Exclusion Criteria:

-

Ages: 1 Day to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 2000-01; Study Completion 2006-12

PRIMARY OUTCOMES:
Diagnostic accuracy

SECONDARY OUTCOMES:
sensitivity, specificity

CONTACTS AND LOCATIONS:
Overall Officials: Shyh-Jye Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - Dept. Medical Imaging, NTUH, Taipei
  - National Taiwan University Hospital, Taipei